CLINICAL TRIAL: NCT00617240
Title: Metformin Mitigation of Atypical Antipsychotic-Induced Metabolic Dysregulation in Adolescent Youth
Brief Title: Strategies to Reduce Antipsychotic-Associated Weight Gain in Youth
Acronym: PREVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 05-2992 GCRC-2501
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Weight Gain
Keywords: antipsychotic; metformin; children; adolescents
MeSH Terms: conditions — Weight Gain | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): metformin in doses from 250mg to 2000mg/day for 26 weeks
  Interventions: Drug: metformin
- 2 (Placebo Comparator): Matched placebo to metformin, doses between 250/0mg and 2000/0mg per day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metformin — 500mg tablets, 250mg to 2000mg/day, po, BID to TID, 26 weeks
  Other Names: Glucophage
  Arms: 1
Drug: placebo — 500/0mg tablets, 250-2000mg/day divided BID to TID, po, 26 weeks
  Arms: 2

SUMMARY:
The purpose of this pilot study is to determine whether starting metformin in conjunction with a second-generation antipsychotic (SGA) and providing information about healthy eating and activity will prevent or reduce the amount of weight gain and the metabolic changes in adolescent youth typically seen with second-generation antipsychotic medication.

DETAILED DESCRIPTION:
This is a 24 week, placebo-controlled, random assignment pilot study in which participants will be randomized in a 1:1 ratio to receive either flexible-dose treatment with metformin for 6 months as well as a newly initiated second generation antipsychotic medication or to receive placebo and the newly initiated antipsychotic medication. All subjects will also be provided healthy lifestyle instruction. The study involves monthly visits for the duration of the study. Participants may be treated as inpatients or outpatients throughout the course of the study. Participants will receive a psychiatric evaluation, physical exam, lab work, ECG, medication treatment, and psychiatric care.

The goal is to evaluate the safety and efficacy of means to prevent and treat weight gain and the associated endocrine, metabolic, and inflammatory changes caused by antipsychotic medications. Behavioral treatments to reduce weight gain and metabolic problems after weight gain has occurred have had little impact. Such interventions must be intensive and sustained over months, if not years to be effective. Although basic lifestyle instruction (diet and physical activity) should be the standard of care for all children and adolescents at risk for becoming overweight, pharmacologic interventions may be the best option for substantially augmenting behavioral approaches to weight management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 10 and 17, male or female, any race or ethnicity
* Any SPMI pediatric diagnosis that meets DSM-IV criteria and frequently is treated with a SGA- typically but not limited to psychotic, mood, pervasive developmental, oppositional defiant, and conduct disorders
* SGA-naïve or less than 2 weeks exposure to any SGA, except ziprasidone
* Legal guardian able and willing to give written informed consent
* If competent, subject able and willing to assent for their own participation

Exclusion Criteria:

* Previous trial of metformin
* Recommendation for treatment with clozapine or ziprasidone
* Current use of insulin or any oral hypoglycemic agent
* Current use of a medication known to mitigate weight gain - amantidine, histamine (H2) antagonists (cimetidine, ranitidine, nizatidine), topiramate, orlistat, sibutramine, stimulants (dextroamphetamine, methylphenidate)
* Any current or past diagnosis of an eating disorder
* Diabetes mellitus
* Current active thyroid (TSH >18 microIU/ml; T4 total >18 mcg/dl), hepatic (2 LFTs >4x upper limits of normal), renal (serum Creatinine >1.4 mg/dL in females and serum Creatinine >1.5 mg/dL in males), cardiac, gastrointestinal, or adrenal disease
* Current substance abuse/dependence within past 2 weeks; a positive urine tox screen at baseline in the absence of meeting criteria for abuse/dependence will not preclude enrollment.
* Pregnancy or breast feeding

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — Unversity of North Carolina, Department of Psychiatry
Locations (1):
- University of North Carolina, Department of Psychiatry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled into the study in January 2007 and enrollment ended in June 2009. All participants came to the ASPIRE clinic for all study visits.
Pre-assignment Details: The study sought to recruit participants who had minimal or no prior exposure to second generation antipsychotics and no previous treatment with metformin.
Groups:
- Metformin: metformin in doses from 250mg to 2000mg/day for 26 weeks
- Placebo: Matched placebo to metformin, doses between 250/0mg and 2000/0,g per day
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.20 (1.643) | 14.25 (2.754) | 14.22 (2.048)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Body Mass Index (BMI)
Description: Change in BMI-Body Mass Index (BMI) is a measure of body fat based on height, weight,gender and chronological age. Change in BMI is calculated as 24 weeks BMI minus the baseline BMI.
Time Frame: 0-24 weeks
Population: All participants who took at least one dose of study treatment and had at least one post baseline assessment.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 5 | 4
kg/m^2 | 1.620 (1.250) | 1.800 (0.5701)

2. Primary Outcome: Change From Baseline to Week 24 in Weight
Description: Change in weight is calculated as 24 weeks weight minus the baseline weight.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 4 | 4
kg | 6.138 (4.346) | 10.45 (5.882)

3. Primary Outcome: Change From Baseline to Week 24 in Fat Mass
Description: Fat mass is a measure of excess body fat. Change in Fat Mass is calculated as 24 weeks fat mass minus the baseline fat mass.
Time Frame: 24 weeks
Population: Only participants with complete data on fat mass at both baseline and 24 weeks were utilized.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 3 | 4
kg | 4.770 (1.770) | 8.225 (1.580)

4. Secondary Outcome: Change From Baseline to Week 24 in Insulin Level
Description: Insulin is a peptide hormone and regulates carbohydrate and fat metabolism in the body.Change in Insulin level is calculated as the 24 weeks insulin level minus the baseline insulin level.
Time Frame: 24 weeks
Population: Only participants with complete data on insulin levels at both baseline and 24 weeks were utilized.
Measure: Mean (Standard Error); unit: microIU/ml
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 2 | 2
microIU/ml | 1.550 (4.250) | 4.80 (2.60)

5. Secondary Outcome: Change From Baseline to Week 24 in Cholesterol Level
Description: According to the lipid hypothesis, abnormal cholesterol levels are strongly associated with cardiovascular disease because these promote atherosclerosis.Cholesterol levels are measured in milligrams (mg) of cholesterol per deciliter(dL) of blood.Change in cholesterol levels is measured at 24 weeks minus the levels at baseline.
Time Frame: 24 weeks
Population: Only participants with complete data on cholesterol levels at both baseline and 24 weeks were utilized.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 4 | 2
mg/dl | -4.250 (17.07) | -31.00 (15.00)

6. Secondary Outcome: Change From Baseline to Week 24 in Triglycerides
Description: In the human body, high levels of triglyceride fats in the bloodstream have been linked to atherosclerosis and, by extension, the risk of heart disease and stroke. A change in triglycerides is calculated from 24 weeks minus baseline levels.
Time Frame: 24 weeks
Population: Only participants with complete data on triglyceride levels at both baseline and 24 weeks were utilized.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 3 | 2
mg/dl | -4.667 (6.766) | -0.5 (0.5)

7. Secondary Outcome: Incidence of Metabolic Syndrome
Description: Metabolic syndrome is a combination of the medical disorders that, when co-occurring, increase the risk of developing cardiovascular disease and diabetes.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 5 | 4
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=5) | Placebo (N=4)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort/pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cold/Flu (Immune system disorders) | 1 (1) | 0 (0)
Respiratory/Ear Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Motor Tics (Nervous system disorders) | 1 (1) | 0 (0)
Low frustration tolerance (Psychiatric disorders) | 1 (1) | 0 (0)
Motor stereotypies (Nervous system disorders) | 1 (1) | 0 (0)
Increased sleep (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed and recruited, however, based on preliminary data, a larger, multi-site trial was developed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No